CLINICAL TRIAL: NCT03112083
Title: Prospective, Randomized, Single-center, Double-blinded, Placebo-controlled Study on Safety and Tolerability of the Krill Powder Product in Slightly Obese Study Subjects With Moderately Elevated Blood Pressure
Brief Title: Safety and Tolerability of Krill Powder Supplement in Slightly Overweight People With Moderately Elevated Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympic Seafood AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: OP001
Record Dates: First submitted 2017-03-27; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Adverse Drug Event; Side Effects of Drugs
Keywords: krill powder; krill oil; safety; tolerability; adverse event; omega-3 fatty acids; eicosapentaenoic acid; docosahexaenoic acid
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: two parallel groups (placebo and Krill oil), intervention trial (56 days)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Krill oil (Active Comparator): Krill powder capsules, 4 g
  Interventions: Dietary Supplement: Nutritional counseling A
- Placebo (Placebo Comparator): Placebo capsules, maize strach, 4 g
  Interventions: Dietary Supplement: Nutritional counselling B

INTERVENTIONS:
Dietary Supplement: Nutritional counseling A — Krill powder capsules
  Arms: Krill oil
Dietary Supplement: Nutritional counselling B — Placebo capsules
  Arms: Placebo

SUMMARY:
The aim of this study was to systematically collect data on safety and tolerability of krill powder in humans and simultaneously gain efficacy data by measuring the risk factors for cardiovascular disease.

The study was a randomised, double-blinded, placebo-controlled intervention study with slightly obese subjects with mildly or moderately elevated blood pressure. Study was conducted at two study sites in Central (Tampere) and Northern Finland (Oulu). In total 35 subjects were randomised according to randomisation list to two groups (krill powder or placebo) in a balanced manner (1:1), separately for both gender and site. Concealed allocation was used to keep both subjects and staff blinded. The study consisted of a pre-screening, Day -7-(-14) screening visit, Day 0 baseline (Randomization visit) and 8-week safety and tolerance follow-up period with three follow-up visits on Day 14, Day 28 and Day 56.

As a primary endpoint of the study, the total number of reported adverse events were compared in the study subject groups taking 8 capsules (4 g) krill oil powder or 8 capsules (4 g) of placebo for the 8-week follow-up period.

DETAILED DESCRIPTION:
Krill powder is a food supplement rich in active ingredients such as fatty acids, phospholipids, protein and antioxidants like astaxanthin. It is considered to be more effective in lowering triglyceride values than fish oils and it may have positive effect on cholesterol values as well. Krill proteins may have positive effect on blood pressure and astaxanthin has anti-oxidative and anti-inflammatory properties. Thus, krill powder has a lot of potential in improving lipid values and having other positive health effects on cardiovascular system. However, there haven't been many clinical studies done with krill powder and thus systematic data on human safety is limited.

The aim of this study was to systematically collect data on safety and tolerability of krill powder in humans and simultaneously gain efficacy data by measuring the risk factors for cardiovascular disease.

The study was a randomised, double-blinded, placebo-controlled intervention study with slightly obese subjects with mildly or moderately elevated blood pressure. Study was conducted at two study sites in Central (Tampere) and Northern Finland (Oulu). In total 35 subjects were randomised according to randomisation list to two groups (krill powder or placebo) in a balanced manner (1:1), separately for both gender and site. Concealed allocation was used to keep both subjects and staff blinded. The study consisted of a pre-screening, Day -7-(-14) screening visit, Day 0 baseline (Randomization visit) and 8-week safety and tolerance follow-up period with three follow-up visits on Day 14, Day 28 and Day 56.

A total of 6 study visits were included. At pre-screening visit the study subjects were requested to sign pre-screening visit informed consent form. A structured interview on demographics (age, sex, ethnicity), previous and current diseases, current medication, alcohol and tobacco consumption and use of dietary supplements (especially fish oil and other n-3 fatty acid (FA) supplements, plant sterols and cholesterol lowering fiber supplements (guar gum, glucomannan, oat fiber etc.) and use of fish foods was carried out at the screening visit and replicated at the day 56 visit. Study included one test product: krill powder derived from antarctic krill (Euphausia Superba) (Rimfrost Pristine®, Rimfrost AS, PO box 234, 6099 Fosnavaag, Norway) and placebo product and both were given in capsule form, 4 capsules in the morning and 4 in the evening.

Nutritional counselling regarding the consumption of fish, omega-3 and -6 fatty acids, food supplements and investigational product for the duration of the study were given for the study subjects at the screening visit by a study nurse or registered dietitian and compliance was followed throughout the study. The subjects were advised to keep their medication, lifestyle, background diet and body weight constant during the study and deviation were recorded into the diary.

As a primary endpoint of the study, the total number of reported adverse events were compared in the study subject groups taking 8 capsules (4 g) krill oil powder or 8 capsules (4 g) of placebo for the 8-week follow-up period. Any unfavourable and unintended sign, symptom or medical complaint and worsening of a pre-existing condition was regarded as adverse event (AE). Study subjects kept diary for the whole duration of the study and were requested to write down all unfavourable symptoms and medical complaints not existing at baseline or significantly worsened from baseline situation. Completeness of diaries was checked at each study visit. All reported adverse events were recorded, coded and analysed carefully to determine severity, possible relation to study products, onset and outcome of the event. In addition, safety laboratory values, cholesterol and triglyceride values and blood pressure was measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Slightly obese female and male subjects (BMI between 25-30 kg/ m2)
* Mildly or moderately elevated blood pressure (RR systolic 130-159/ diastolic under 99)
* Signed written informed consent

Exclusion Criteria:

* Medication potential to affect serum lipids (lipid-lowering drugs)
* Familial hypercholesterolemia, marked combined hyperlipidemia, condition that would impair fat absorption (e.g. chronic pancreatitis, pancreatic lipase deficiency syndrome)
* Any untreated medical condition affecting absorption of fat
* Type 1 and 2 diabetes
* Cancer or other malignant disease within the past five years
* Periodical hormone replacement therapy
* High intake of oily fish (>2 times per week as a principal meal) (i.e. salmon, herring, sardines, mackerel, vendace)
* Smoking
* Alcohol consumption >15 doses per week
* Pregnant, lactating or wish to become pregnant
* Hypersensitivity to fish or any of the components of the test products
* Regular use (> 3 times per week) of n-3 or other fatty acid supplements, plant sterols or fiber supplements 4 weeks before randomization
* Lack of suitability for participation in the trial, for any medical reason, as judged by the PI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2016-06-17 (Actual)

PRIMARY OUTCOMES:
Change in Adverse events | Screening, baseline, day 28, day 56
  Total number of reported adverse events

SECONDARY OUTCOMES:
Type of adverse event | Screening, baseline, day 28, day 56
  Coding by MedDRA and reported with System organ class (SOC) and Prefered term (PT) levels, seriousness, severity, onset and causality of the reported adverse events
Change in Systolic blood pressure | Screening, baseline, day 28, day 56
  Mean and mean change (0 vs 8 wk) in systolic blood pressure recorded with 1 mmHg accuracy taken in the screening and during the intervention visits (three measurements are taken altogether and an average of last two measures is used in the analysis)
Change in Diastolic blood pressure | Screening, baseline, day 28, day 56
  Mean and mean change (0 vs 8 wk) in diastolic blood pressure recorded with 1 mmHg accuracy taken in the screening and during the intervention visits (three measurements are taken altogether and an average of last two measures is used in the analysis)
Change in thyrotropin | Screening, baseline, day 28, day 56
  Regular safety parameters from the blood including mean and median variables of blood thyrotropin
Change in Alanine transaminase (ALT) | Screening, baseline, day 28, day 56
  Regular safety parameters from the blood including mean and median variables of blood Alanine transaminase (ALAT)
Change in Aspartate transaminase (AST) | Screening, baseline, day 28, day 56
  Regular safety parameters from the blood including mean and median variables of blood Aspartate transaminase (ASAT)
Change in blood glucose | Screening, baseline, day 28, day 56
  Regular safety parameters from the blood including mean and median variables of blood glucose
Change in gamma glutamyl transferase | Screening, baseline, day 28, day 56
  Regular safety parameters from the blood including mean and median variables of gamma glutamyl transferase
Change in creatinine | Screening, baseline, day 28, day 56
  Regular safety parameters from the blood including mean and median variables of creatinine
Change in blood count | Screening, baseline, day 28, day 56
  Regular safety parameters from the blood including mean and median variables of blood count
Change in Thyroid stimulating hormone (TSH) | Screening, baseline, day 28, day 56
  Regular safety parameters from the blood including mean and median variables of Thyroid stimulating hormone (TSH)
Change in Triglycerides | Screening, baseline, day 28, day 56
  Mean concentration of serum total triglycerides and mean change (0 vs 8 wk) in serum total and lipoprotein lipids
Change in total cholesterol | Screening, baseline, day 28, day 56
  Mean concentration of total cholesterol during the 8-week intervention and mean change (0 vs 8 wk) in serum total and lipoprotein lipids
Change in Low density lipoproteine (LDL)-cholesterol | Screening, baseline, day 28, day 56
  Mean concentration of serum LDL-cholesterol during the 8-week intervention and mean change (0 vs 8 wk) in serum total and lipoprotein lipids
Change in High density lipoproteine (HDL)-cholesterol | Screening, baseline, day 28, day 56
  Mean concentration of serum HDL-cholesterol during the 8-week intervention and mean change (0 vs 8 wk) in serum total and lipoprotein lipids

CONTACTS AND LOCATIONS:
Locations (1):
- Oy Medfiles Ltd, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarkkinen ES, Savolainen MJ, Taurio J, Marvola T, Bruheim I. Prospective, randomized, double-blinded, placebo-controlled study on safety and tolerability of the krill powder product in overweight subjects with moderately elevated blood pressure. Lipids Health Dis. 2018 Dec 20;17(1):287. doi: 10.1186/s12944-018-0935-x. PMID 30572894